CLINICAL TRIAL: NCT06893211
Title: Effect of Tirzepatide-Induced Weight Loss on Adipose Tissue in Obesity
Brief Title: Effect of Tirzepatide on Brown Adipose Tissue in Obesity
Acronym: TABFAT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0120-56/2024-2711-7
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Obesity
Keywords: obesity; tirzepatide; brown adipose tissue; beige adipose tissue; adipose tissue browning; energy expenditure
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tirzepatide (Experimental)
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide is a dual glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide-1 (GLP-1) receptor agonist. It will be administered via subcutaneous injection once weekly in a dose-titration scheme: starting at 2.5 mg, and increased every 4 weeks by 2.5 mg up to a maximum of 15 mg, based on tolerability. The medication will be supplied in prefilled pens identical in appearance to placebo pens.
  Arms: Tirzepatide
Drug: Placebo — Placebo will be administered via subcutaneous injection once weekly using pens that are visually indistinguishable from those used for tirzepatide. Dose escalation will follow the same schedule (2.5 mg-equivalent increments every 4 weeks) to preserve blinding integrity.
  Arms: Placebo

SUMMARY:
This study is testing whether a new anti-obesity medicine called tirzepatide can increase the activity of special fat cells in the body that help burn energy. These fat cells are known as brown and beige fat. The study includes women with obesity and will last 24 weeks.

Participants will receive either tirzepatide or a placebo (a look-alike injection with no active drug). Researchers will measure the amount and activity of brown fat using medical imaging (PET/CT, MRI, and thermal camera), and examine fat tissue samples to look for changes in gene activity and structure that show beige fat activation.

The study will also evaluate how these fat changes affect body weight, energy use, hormone levels, blood sugar, and other health markers. The goal is to learn whether tirzepatide helps improve metabolism by increasing energy-burning fat in addition to reducing appetite.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age between 18 and 50 years
* BMI between 30 kg/m² and 40 kg/m² at pre-screening
* Prior comprehensive non-pharmacological and non-surgical management of obesity, including a history of at least 12 months of intensive lifestyle intervention with a maximum weight reduction of less than 5%
* Stable body weight within the three months preceding study enrollment (defined as weight fluctuations within 5%)
* No prior pharmacological or surgical interventions for obesity
* Euthyroid state
* Eumenorrhea or Oligomenorrhea
* Ability to comprehend the study objectives and procedures
* Willingness to provide informed consent and to comply with the study protocol, including the use of highly effective contraception during the study period, with signed consent and agreement provided in duplicate
* Commitment to use highly reliable contraception and absence of plans for pregnancy within the 8 months following enrollment

Exclusion Criteria:

* Pregnancy or lactation
* Postmenopausal
* Amenorea
* Type 2 diabetes
* Reliance on natural contraception methods
* Non-compliance with previous therapeutic regimens
* Personal history of malignancy
* Personal or family history of medullary thyroid carcinoma
* Personal history of pancreatitis
* Personal history of cholelithiasis
* Personal history of major depressive episodes or suicidal ideation
* Personal history of acute coronary events or hemodynamically significant coronary artery disease
* Psychiatric disorders
* Current treatment with sympathomimetics or sympatholytics
* Excessive alcohol consumption

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Brown Adipose Tissue Activity and Volume | Baseline to Week 24
  Assessed using 18F-FDG-PET/CT, magnetic resonance imaging (MRI), and infrared thermography. Outcome measured as change in mean standardized uptake value, supraclavicular skin temperature, and BAT volume in predefined anatomical regions (supraclavicular and cervical areas) between baseline and after 24 weeks of treatment.
Change in Molecular Markers of Browning in Subcutaneous White Adipose Tissue | Baseline to Week 24
  Measured as changes in the expression levels of uncoupling protein 1 (UCP1) and other browning-associated genes (via RT-PCR and RNA sequencing) in subcutaneous white adipose tissue (WAT) biopsies. Additionally, assessed through histomorphometric analysis of adipocyte phenotype, including the proportion of multilocular (plurivacuolar) adipocytes, immune cell infiltration, and microvascular density, to characterize tissue remodeling indicative of beige adipocyte induction.

SECONDARY OUTCOMES:
Correlation Between Different BAT Assessment Methods | Baseline and Week 24
  Comparative analysis between 18F-FDG-PET/CT, MRI fat fraction, and infrared thermography for assessing BAT activity and volume.
Change in Resting Energy Expenditure | Baseline to Week 24
  Measured by indirect calorimetry using a portable metabolic analyzer. Outcome reported as absolute change in REE (kcal/day).
Association Between Changes in Resting Energy Expenditure, Metabolic Health Markers, and Thermogenic Adipose Tissue | Baseline to Week 24
  Assessed by evaluating correlations between changes in resting energy expenditure (REE, measured by indirect calorimetry), metabolic health parameters (including glucose metabolism, insulin sensitivity indices, lipid profile, and hormonal markers), body composition changes, and alterations in thermogenic adipose tissue activity and volume (as measured by 18F-FDG-PET/CT, MRI, and thermography). This outcome aims to determine the interrelationship between metabolic adaptations and thermogenic fat activation following tirzepatide treatment.
Association Between Resting Energy Expenditure, Metabolic Health Markers, and Thermogenic Adipose Tissue | Baseline
  Assessed by evaluating correlations between anthropometric data, resting energy expenditure (REE, measured by indirect calorimetry), metabolic health parameters (including glucose metabolism, insulin sensitivity indices, lipid profile, and hormonal markers), body composition, and thermogenic adipose tissue activity and volume (as measured by 18F-FDG-PET/CT, MRI, and thermography). This outcome aims to determine variables that correlate with pre-treatment thermogenic adipose tissue quantity and activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Diabetes and Metabolic Diseases, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) to be shared will include demographic data, basic clinical measurements, body composition assessment, laboratory results, imaging data, resting energy expenditure measurements, molecular data and histological features from subcutaneous adipose tissue biopsies. All shared data will be fully de-identified, and no directly identifiable personal information will be included.

REFERENCES:
- [Derived] Herman R, Jensterle M, Horvat S, Lezaic L, Snoj Z, Pusnik I, Goricar K, Cor A, Pusnik L, Mlacnik V, Hanzelic L, Janez A. Effect of tirzepatide-induced weight loss on adipose tissue in obesity: rationale and design of the randomized placebo-controlled Tirzepatide Brown and Beige Adipose Tissue Activation (TABFAT) trial. Trials. 2025 Aug 22;26(1):300. doi: 10.1186/s13063-025-09045-9. PMID 40847412